CLINICAL TRIAL: NCT01221844
Title: Phase IV Study of Oral Administration of Bovine Lactoferrin (bLf) to Prevent and Cure Iron Deficiency (ID) and Iron Deficiency Anemia (IDA) Until Delivery in Hereditary Thrombophilia (HT) Affected Pregnant Women
Brief Title: Bovine Lactoferrin to Prevent and Cure Iron Deficiency and Iron Deficiency Anemia in Complicated Pregnancies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clinica Fabia Mater (Other)
Responsible Party: Dr Rosalba Paesano, Clinica Fabia Mater, Rome (Italy)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RP2010
Record Dates: First submitted 2010-10-12; First posted 2010-10-15 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Pregnancy; Iron Deficiency; Iron Deficiency Anemia
Keywords: Lactoferrin; Pregnancy; Hereditary Thrombophilia; Iron deficiency; Iron deficiency anemia
MeSH Terms: conditions — Iron Deficiencies; Anemia, Iron-Deficiency; Thrombophilia, hereditary | interventions — ferrous sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactoferrin treatment in HT pregnacies (Experimental): Pregnant women affected by HT, ID and IDA are enrolled and treated until delivery with oral administration of one capsule of 100 mg of bLf (Lattoglobina, Grunenthal, Italy) twice a day before meals. In twin pregnancies or in severe anemia, HT pregnant women are treated until delivery with two capsules of 100 mg of bLf twice a day, before meals.
  Interventions: Dietary Supplement: Lattoglobina (Grunenthal) containing bLf
- Ferrous sulfate in HT pregnancies (Active Comparator): Pregnant women affected by HT, ID and IDA are enrolled and treated until delivery with oral administration of 520 mg of ferrous sulfate (Ferro-Grad, Abbott Laboratories, USA), once a day during meal.
  Interventions: Drug: FerroGrad by Abbott

INTERVENTIONS:
Dietary Supplement: Lattoglobina (Grunenthal) containing bLf — One capsule of Lattoglobina contains 100 mg of bLf. Dosage: one capsule twice a day before meals. In twin pregnancy or in severe anemia the dosage is increased to 2 capsules twice a day before meals
  Other Names: Commercialization by Grunenthal Italy; Manifacture by Giellepi; Licence Microbo srl, Rome, Italy
  Arms: Lactoferrin treatment in HT pregnacies
Drug: FerroGrad by Abbott — Dosage: one tablet/day containing 540 mg of ferrous sulfate during meals
  Other Names: FerroGrad; Abbott
  Arms: Ferrous sulfate in HT pregnancies

SUMMARY:
The purpose of this study is to determine whether bovine lactoferrin is effective in preventing and curing iron deficiency and iron deficiency anemia in Hereditary Thrombophilia affected women during pregnancy.

The proposed clinical trial is considered as PHASE IV because in Italy bLf is commercialized by Grunenthal, as Lattoglobina® (capsules with 100 mg of bLf), to prevent and cure iron deficiency and iron deficiency anemia in pregnant women.

DETAILED DESCRIPTION:
In industrialized and developing countries, iron deficiency (ID) and iron deficiency anemia (IDA) are highly prevalent in pregnant women. ID and IDA, in pregnant women as a consequence of an increased iron requirement, due to enhanced blood volume and development of fetal-placenta unit, represent a high risk for maternal and infant health: preterm delivery, fetal growth retardation, low birth weight, and inferior neonatal health. However, the degree of fetal ID is not always as severe as that in mother, being iron transfer from the mother to the fetus regulated by the placenta. In particular, the placental syncytiotrophoblast acquires ferric iron bound to maternal transferrin at the apical membrane through transferrin receptors (TfR-1), which noticeably increase in pregnant women suffering of ID and IDA. Recently, it has been suggested that most iron transfer to the fetus, occurring after the 30th week of gestation, also involves placental expression of hepcidin and ferroportin, two proteins known to modulate systemic iron homeostasis in adults. As matter of fact, iron homeostasis is tightly regulated through iron absorption, storage and transport. The absorption of nearly all dietary iron (1-2 mg daily), ensuring iron supplies in the bone marrow, at second and third trimester of pregnancy increases until to about 4 and 8 mg/day, respectively. The iron absorption takes place in the proximal duodenum and includes the following steps: (i) reduction of iron from the ferric state (III) to the ferrous state (II) by a ferrireductase (duodenal cytochrome B; (ii) apical uptake by enterocytes followed by trans-cellular trafficking via divalent metal transporter 1; (iii) storage into ferritin; and (iv) basolateral efflux by the iron transporter ferroportin. Ferroportin, the only known cellular iron exporter from tissues into blood, has been found in all cell types involved in iron export, including the enterocytes, hepatocytes, placental cells and macrophages which require ferroportin to daily recycle 20 mg of iron from lysed erythrocytes for erythropoiesis.

Another pivotal component of systemic iron homeostasis is hepcidin, a circulating peptide hormone synthesized by hepatocytes in iron loading conditions and secreted in plasma and urine. Hepcidin regulates the entry of iron into plasma through ferroportin. Hepcidin, by binding to ferroportin, causes ferroportin phosphorylation, internalization and degradation in lysosomes, thus hindering iron export and enhancing cytosolic iron storage in ferritin. Iron homeostasis disorders appear to arise from hepcidin and/or ferroportin dysregulation. Similarly to the regulation of maternal systemic iron homeostasis, fetal hepcidin controls the transfer of maternal iron across the placenta to the fetus and the enhanced placental-fetal iron transport is related to an increased expression of ferroportin on placental basal fetal-facing membrane, consistent with unidirectional mother-fetus iron transport. Even if the interaction of hepcidin with ferroportin can explain the regulation of iron homeostasis at systemic level, the influence of iron metabolism on critical stage of fetal development, is still unknown.

Regulation of hepcidin expression seems to occur at transcriptional level and its production is increased by iron loading and inflammation and decreased by anemia and hypoxia.

Even if the molecular mechanisms of hepcidin regulation by iron, oxygen and anemia are still unclear, it is known that Interleukin 6 (IL-6) induces transcription of the hepcidin gene in hepatocytes. In inflammatory and infection disorders, cytokine induced hepcidin excess, through ferroportin binding, contributes to development of anemia of inflammation, characterized by ID and IDA despite adequate iron stores. When iron export is hindered, iron is stored in host cells. However, inflammation may contribute to ID and IDA by hepcidin-independent mechanism(s) as the down-regulation of ferroportin. Independently on hepcidin synthesis, high levels of serum IL-6 seem to down-regulate ferroportin mRNA expression, thus sequestering iron inside cells and blocking iron flow into plasma. The inability to export iron leads to hypoferremia, decreased pool of serum transferrin-Fe(III) and iron-limited erythropoiesis.

The recent discovery of hepcidin-ferroportin complex has greatly contributed to clarify the enigmatic mechanism of systemic iron homeostasis. Notwithstanding, iron homeostasis disorders, as ID and IDA, are still treated with oral administration of large quantity of iron as fer¬rous sulfate due to its poor bio-availability. Ferrous sulfate oral administration often fails to exert significant effects on ID and IDA, and frequently causes many adverse effects, including gastrointestinal discomfort, nausea, vomiting, diarrhea, and constipation.

Recently, a significant decrease of total serum iron and serum ferritin concentrations related with an increase of serum IL-6 concentration has been observed in pregnant women and in hemodialysis patients, orally treated with ferrous sulfate. Therefore, it can be hypothesized that supplemented iron was not exported from cells to circulation, but it was accumulated inside the cells, thereby increasing inflammatory status, similarly to that reported in animals treated with ferrous sulfate.

The weight of evidences, which let to doubt on the efficacy and safety of ferrous sulfate oral administration, has stimulated the research of more effective approaches to prevent ID and toxicity associated with iron overload. The treatment of ID and IDA during pregnancy should be entirely reconsidered taking into account not only the enhanced blood volume and development of fetal-placenta unit, but also other factors, as IL-6, which, inducing hepcidin up-regulation and ferroportin down-regulation, can play a pivotal role in iron homeostasis disorders.

For this purpose, lactoferrin (Lf), a cationic iron-binding glycoprotein, able to chelate at high affinity (KD w10/20 M) two ferric ions per molecule (30), is emerging as an important regulator of systemic iron homeostasis, able to cure ID and IDA. Lf is synthesized by exocrine glands and neutrophils in infection and inflammation sites. In humans, free iron does not exceed 10-18 M to avoid precipitation, microbial growth and formation of reactive oxygen species. Lf in tissues and secretions and transferrin in blood assure that iron was bound and scarcely available as free-ion.

Even if several functions, dependent and independent on its iron binding ability, have been attributed to Lf, our recent clinical trials have demonstrated that this natural compound may represent an interesting approach in the therapy for ID and IDA in pregnant women. As matter of fact, a milk derivative bovine lactoferrin (bLf) restores the physiological transport of iron from tissues to circulation, thus curing ID and IDA. Moreover, differently from ferrous sulfate, bLf oral administration exerts an anti-inflammatory effect by decreasing serum IL-6 concentration in uncomplicated pregnancies.

The hypercoagulable state represents one of the physiological changes occurring during pregnancy. The hereditary thrombophilia (HT), a genetic predisposition to inappropriately form clots, significantly increases adverse outcomes including recurrent miscarriages, intrauterine fetal death and growth retardation, preeclampsia and placental abruption. It is well known that inflammation promotes coagulation and IL-6 high levels in plasma of HT affecting pregnant women with severe preeclampsia have been found. Moreover, elevated intra-amniotic IL-6 and IL-8 levels have been correlated to preterm birth.

Therefore, iron supplementation via oral administration of ferrous sulfate increasing serum IL-6 levels in uncomplicated pregnancies, could be deleterious in HT affecting pregnant women and could contribute to enhance iron overload in tissues, inflammation and cell damages.

The bLf capability to prevent and cure ID and IDA together with its ability of decreasing serum IL-6 concentration could be effective even in the treatment of ID and IDA in pregnant women affected by HT.

In this clinical trial, pregnant women affected by hereditary thrombophilia (HT), suffering of ID and IDA, receive an oral administration of bovine Lf (bLf) 100 mg/twice a day or ferrous sulfate 520 mg/day. The number of red blood cells, the values of hemoglobin, total serum iron, serum ferritin, haematocrit, serum Interleukin-6 (IL-6) and prohepcidin are assayed before therapy, every 30 days until delivery.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with one of genetic thrombophilia markers as factor V Leiden, prothrombin 20210A mutation, antiphospholipid antibodies, hyperhomocysteinemia and deficiencies of antithrombin, protein C, or protein S.
* pregnant women affected by HT and suffering of iron deficiency (ID) and iron deficiency anemia (IDA)
* different trimester of pregnancy
* previous miscarriage/s
* previous preterm delivery/ies
* iron disorders as iron deficiency and iron deficiency anemia are defined by the number of red blood cells <4.000.000/mL, the hemoglobin concentration ≤ 11 g/dL, the total serum iron ≤ 30 mg/dL and serum ferritin ≤12 ng/mL.

Exclusion Criteria:

* absence of iron deficiency and iron deficiency anemia
* non-pregnant women
* uncomplicated pregnancies
* no informed consent
* other treatments of iron supplementation
* recent blood transfusion
* other concomitant diseases
* ascertained allergy to milk proteins or to iron products.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Hematological parameters | At time 0 (enrollement) and every 30 days until delivery (6-8 months)
  Efficacy of bLf versus ferrous sulfate in preventing and curing iron deficiency and iron deficiency anemia

SECONDARY OUTCOMES:
Side effects | 6-8 months
  Control of side effects of oral administration of bLf and ferrous sulfate as:
  * gastrointestinal discomfort
  * nausea
  * vomiting
  * diarrhea
  * constipation

CONTACTS AND LOCATIONS:
Overall Officials: Rosalba Paesano, Dr, Study Chair — Clinica Fabia Mater, Via Olevano Romano 25, Rome (Italy)
Locations (1):
- Clinica Fabia Mater, Rome, Rm, Italy

REFERENCES:
- [Background] Paesano R, Berlutti F, Pietropaoli M, Goolsbee W, Pacifici E, Valenti P. Lactoferrin efficacy versus ferrous sulfate in curing iron disorders in pregnant and non-pregnant women. Int J Immunopathol Pharmacol. 2010 Apr-Jun;23(2):577-87. doi: 10.1177/039463201002300220. PMID 20646353
- [Background] Paesano R, Berlutti F, Pietropaoli M, Pantanella F, Pacifici E, Goolsbee W, Valenti P. Lactoferrin efficacy versus ferrous sulfate in curing iron deficiency and iron deficiency anemia in pregnant women. Biometals. 2010 Jun;23(3):411-7. doi: 10.1007/s10534-010-9335-z. Epub 2010 Apr 21. PMID 20407805
- [Background] Paesano R, Pietropaoli M, Gessani S, Valenti P. The influence of lactoferrin, orally administered, on systemic iron homeostasis in pregnant women suffering of iron deficiency and iron deficiency anaemia. Biochimie. 2009 Jan;91(1):44-51. doi: 10.1016/j.biochi.2008.06.004. Epub 2008 Jun 14. PMID 18601971
- [Background] Paesano R, Torcia F, Berlutti F, Pacifici E, Ebano V, Moscarini M, Valenti P. Oral administration of lactoferrin increases hemoglobin and total serum iron in pregnant women. Biochem Cell Biol. 2006 Jun;84(3):377-80. doi: 10.1139/o06-040. PMID 16936810
- [Derived] Lepanto MS, Rosa L, Cutone A, Conte MP, Paesano R, Valenti P. Efficacy of Lactoferrin Oral Administration in the Treatment of Anemia and Anemia of Inflammation in Pregnant and Non-pregnant Women: An Interventional Study. Front Immunol. 2018 Sep 21;9:2123. doi: 10.3389/fimmu.2018.02123. eCollection 2018. PMID 30298070
- [Derived] Paesano R, Pacifici E, Benedetti S, Berlutti F, Frioni A, Polimeni A, Valenti P. Safety and efficacy of lactoferrin versus ferrous sulphate in curing iron deficiency and iron deficiency anaemia in hereditary thrombophilia pregnant women: an interventional study. Biometals. 2014 Oct;27(5):999-1006. doi: 10.1007/s10534-014-9723-x. Epub 2014 Mar 4. PMID 24590680